CLINICAL TRIAL: NCT06328712
Title: An Open, Dose-escalation, Phase 1b Clinical Trial to Evaluate the Safety and Efficacy of EN001 in Patients With Charcot-Marie-Tooth Disease Type 1A (CMT1A)
Brief Title: Evaluate the Safety and Efficacy of EN001 in Patients With Charcot-Marie-Tooth Disease Type 1A
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ENCell (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EN001_MIRACLE1
Record Dates: First submitted 2024-02-19; First posted 2024-03-25 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Charcot-Marie-Tooth Disease Type 1A
MeSH Terms: conditions — Charcot-Marie-Tooth Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Active Comparator): EN001 1.25×10^6 cells/kg
  Interventions: Drug: EN001
- Cohort 2 (Active Comparator): EN001 2.5×10^6 cells/kg
  Interventions: Drug: EN001

INTERVENTIONS:
Drug: EN001 — * Cohort 1: EN001 1.25×10^6 cells/kg administered intravenously (IV) 2 times at 4 week intervals.
  * Cohort 2: EN001 2.5×10^6 cells/kg administered intravenously (IV) 2 times at 4 week intervals.
  Other Names: EN001(Allogeneic early-passage Wharton's jelly-derived mesenchymal stem cells(WJ-MSCs) )

SUMMARY:
An Open, Dose-escalation, Phase 1b Clinical Trial to Evaluate the Safety and Efficacy of EN001 in Patients with Charcot-Marie-Tooth Disease type 1A (CMT1A)

DETAILED DESCRIPTION:
This clinical trial is a phase 1b clinical trial with a 3+3 dose escalation design to evaluate the safety, including tolerability, of EN001 and explore efficacy.

The study was designed using the traditional 3+3 dose escalation method to confirm the maximum tolerated dose (MTD) and determine the recommended phase 2 dose (RP2D).

Dose increase is carried out until the maximum tolerated dose (MTD) is confirmed at a dose of 2.5 × 10^6 cells/kg (Cohort 2) or less, which is the maximum planned dose (MPD). The maximum tolerated dose (MTD) is defined as the highest dose at which the incidence of dose limiting toxicity (DLT) is lower than 33%. To determine the maximum tolerated dose (MTD), 3-6 test subjects from each dose cohort are enrolled and EN001 is administered twice at 4-week intervals, and dose-limiting toxicity (DLT) is evaluated until 4 weeks (visit 6).

The safety review committee (SRC) is comprised of the principal investigator, sponsor, etc. as members, and EN001 confirmed by the end of each cohort (end of dose-limiting toxicity (DLT) evaluation of the last dosed subject in the cohort). Safety data are comprehensively reviewed to determine all matters related to dose, such as increase or decrease in dose, and finally the recommended phase 2 dose (RP2D) is determined.

In addition, test subjects participating in phase 1b will be followed up for safety and effectiveness for 5 years from the time of EN001 administration according to the long-term follow-up protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who have voluntarily agreed to participate in this clinical trial.
2. Men and women aged 19 years or older at the time of providing written consent.
3. Individuals who meet all of the following genetic and clinical diagnostic criteria:

   1. Genetic diagnosis: CMT1A type
   2. Clinical diagnosis:

      * Those with a CMT Neuropathy Score version 2 (CMTNSv2) between 2 or more and 20 or less.
      * Those experiencing muscle weakness due to foot dorsiflexion impairment.
4. Women and men of childbearing potential who have agreed to use the appropriate contraceptive method(s) outlined in the protocol during the clinical trial period.

   * Appropriate contraception is defined as follows and is achieved by applying one or more methods of contraception.

     * Hormonal contraceptives
     * Implantation of an intrauterine device or intrauterine system
     * Sterilization procedures (vasectomy, tubal ligation, etc.)
     * Double contraceptive method: male condom along with other contraceptive methods [hormonal contraceptives (oral contraceptives, subcutaneous contraceptives (Implanon, etc.), long-acting contraceptive injections, emergency contraceptive pills), implantation of an intrauterine device or intrauterine system (Loop, Mirena), Infertility procedures (vasectomy, tubal ligation, etc.)]
     * Abstinence: Absolute abstinence. If, in the examiner's judgment, the subject's age, occupation, lifestyle, or sexual orientation warrants contraception, strict abstinence from sexual intercourse is also acceptable. However, periodic abstinence (e.g. Karenda method, ovulation method, symptomatic temperature method), abstinence, and external vaginal ejaculation are not recognized as appropriate contraceptive methods.

Exclusion Criteria:

1. Those with the following comorbidities confirmed at the time of screening

   1. Subjects with neuromuscular diseases other than CMT1A or neuropathy- inducing factors (uremia) that may affect the safety and efficacy evaluation of this clinical trial, according to the judgment of the investigator.
   2. Individuals diagnosed with type 1 or type 2 diabetes
   3. Individuals diagnosed with active pulmonary tuberculosis
   4. Patients with uncontrolled hypertension (systolic blood pressure over 180 mmHg or diastolic blood pressure over 110 mmHg)
   5. Subjects with other clinically significant diseases, including significant heart, lung, liver, kidney, hematological, immunological or behavioral diseases or malignant tumors, according to the investigator's judgment
   6. Individuals who display the specified test abnormalities in laboratory tests at the time of screening:

      * AST or ALT > 3 x ULN
      * Total bilirubin> 1.5 x ULN
      * Serum creatinine > 1.5 x ULN
      * Any one of the serum virus tests (HBsAg, anti-HBc, anti-HCV, HIV Ag/Ab) is positive (If anti-HBc positive) However, registration is possible if the HBV DNA test result is negative. (If anti-HCV positive) However, registration is possible if the HCV RNA test result is negative.
   7. Those who have ankle contracture or have undergone surgery that may affect muscle strength measurement tests
2. Medical history and surgical history

   1. Those who have undergone orthopedic surgery (bone or ligament correction, artificial joint implantation, osteotomy, arthroscopic surgery) on the lower extremities within 24 weeks before screening
   2. Those with a history of stroke or cerebral ischemic attack within 48 weeks before screening
   3. Those with a history of coronary artery disease, such as myocardial infarction or incomplete angina, within 48 weeks before screening
   4. Those with a history of malignant tumor within 240 weeks before screening (excluding basal cell carcinoma or squamous cell carcinoma that occurs on the skin)
3. Drugs and therapies prohibited from concurrent use

   1. Those who participated in another clinical trial and administered/applied clinical trial drugs/medical devices within 4 weeks before screening
   2. Those who administered/applied immunosuppressants, chemotherapy, radiation therapy, etc. within 12 weeks before screening
   3. Persons who have administered cell therapy or gene therapy throughout their lives
   4. Persons who have administered neurotoxic drugs that can accelerate peripheral nerve damage

      * Platinum series: cisplatin, carboplatin, oxaliplatin
      * Taxane series: paclitaxel, docetaxel
      * Proteasome inhibitors: bortezomib, carfilzomib, ixazomib, etc.
      * thalidomide and derivatives: thalidomide, lenalidomide, pomalidomide
      * Vinca alkaloid series: vincristine, vinblastine, vindesine, vinorelbine
      * Antiarrhythmic drug: amiodarone
      * Anti-inflammatory and antibiotic: colchicine, nitrofurantoin
      * Antiretroviral drugs: zalcitabine, stavudine
      * Others: dichloroacetate, tacrolimus, suramin
4. Persons with hypersensitivity to the components of clinical investigational products
5. Those who have had metal substances (heart pacemaker, nerve stimulator, cochlear implant, etc.) implanted in their body
6. Pregnant, lactating, or planning to become pregnant during the clinical trial period
7. Subjects with a psychiatric disorder (anxiety disorder, claustrophobia, or other significant mental disorder) or a history of drug and alcohol abuse that may affect the clinical trial, according to the judgment of the investigator.
8. Those who are deemed inappropriate to participate in clinical trials according to the judgment of the investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) and adverse drug reactions related to discontinuation of investigational product administration | Up to 8 weeks
  Present the frequency and percentage of dose-limiting toxicity (DLT) occurrence across dose cohorts, along with detailed information on the types of DLTs.
  Adverse events related to discontinuation of clinical investigational drug administration, discontinuation of clinical investigational drug administration Regarding related adverse drug reactions, the number of subjects in each cohort, incidence rate (%), and Two-sided 95% confidence intervals and number of occurrences are presented.

SECONDARY OUTCOMES:
CMTNSv2 score change | At 4, 8, 18, and 24 weeks compared to baseline (Visit 2)
  Present the subject count, mean, standard deviation, median, minimum, and maximum for the changes at each time point within each dosage group.
CMT examination score change | At 4, 8, 18, and 24 weeks compared to baseline (Visit 2)
  Present the subject count, mean, standard deviation, median, minimum, and maximum for the changes at each time point within each dosage group.
Rasch-modified CMTNSv2 score change | At 4, 8, 18, and 24 weeks compared to baseline (Visit 2)
  Present the subject count, mean, standard deviation, median, minimum, and maximum for the changes at each time point within each dosage group.
Rasch-modified CMTES score change | At 4, 8, 18, and 24 weeks compared to baseline (Visit 2)
  Present the subject count, mean, standard deviation, median, minimum, and maximum for the changes at each time point within each dosage group.
FDS score change | At 4, 8, 18, and 24 weeks compared to baseline (Visit 2)
  Present the subject count, mean, standard deviation, median, minimum, and maximum for the changes at each time point within each dosage group.
ONLS score change | At 4, 8, 18, and 24 weeks compared to baseline (Visit 2)
  Present the subject count, mean, standard deviation, median, minimum, and maximum for the changes at each time point within each dosage group.
10MWT score change | At 4, 8, 18, and 24 weeks compared to baseline (Visit 2)
  Present the subject count, mean, standard deviation, median, minimum, and maximum for the changes at each time point within each dosage group.
Change in grade of fatty infiltration in the proximal lower extremities (According to Goutallier classification scale) | At 24 weeks compared to baseline (Visit 2)
  Present the subject count, mean, standard deviation, median, minimum, and maximum for the changes at each time point within each dosage group.
Change in Motor Nerve Conduction Velocity (Unit: m/s) | At 4, 8, 18, and 24 weeks compared to baseline (Visit 2)
  Present the subject count, mean, standard deviation, median, minimum, and maximum for the changes at each time point within each dosage group.
Change in Compound Muscle Action Potential (Unit: ㎷) | At 4, 8, 18, and 24 weeks compared to baseline (Visit 2)
  Present the subject count, mean, standard deviation, median, minimum, and maximum for the changes at each time point within each dosage group.
Change in Sensory Nerve Action Potential (Unit: ㎶) | At 4, 8, 18, and 24 weeks compared to baseline (Visit 2)
  Present the subject count, mean, standard deviation, median, minimum, and maximum for the changes at each time point within each dosage group.
Change in Sensory Nerve Conduction Velocity (Unit: m/s) | At 4, 8, 18, and 24 weeks compared to baseline (Visit 2)
  Present the subject count, mean, standard deviation, median, minimum, and maximum for the changes at each time point within each dosage group.
SF-36v2 score change | At 24 weeks compared to baseline (Visit 2)
  Present the subject count, mean, standard deviation, median, minimum, and maximum for the changes at each time point within each dosage group.
Adverse Event | Up to 24weeks. However, adverse drug reactions that persist at the end of the clinical trial will be followed up until the possible adverse reactions are resolved or it is determined that further follow-up is not meaningful.
  By cohort that Number of subjects, incidence rate (%), confidence interval (two-sided 95%), presents the number of occurrences. Additional, The pre-treatment adverse event that occurred before administration of clinical trial drugs is presented in detail.
Vital sign | Up to 24 weeks
  Number of participants with clinically significant abnomalities in vital signs after EN001 administration.
  Vital Signs include blood pressure (mmHg), pulse (times/minute), respiratory rate (times/minute), and body temperature (℃) and will be assessed.
  By cohort and visit, present continuous variables with subject count, mean, standard deviation, median, minimum, and maximum. For categorical variables, provide shift table.
Laboratory examination | Up to 24 week. Serum virus testing is performed only during screening. At Baseline and Week 4, hematological tests, blood chemical tests, TCO2, Mg, and blood coagulation tests are performed before and within 4 hours after administration of the IP.
  Number of participants with clinically significant abnormalities in Laboratory parameters after EN001 administration.
  Hematological tests, Blood chemical tests, Blood coagulation test, Urine test, Serum virus test.
  It is conducted through blood and urine collection, and the PI checks whether the test results are normal, abnormal, and clinically significant.
electrocardiography | At Baseline, Week 4, Week 8, Week 12, Week 18, Week 24
  Number of participants with clinically significant abnormalities in electrocardiography after EN001 administration.
  Based on the PR Interval, QRS Duration, QTc Interval and QTcF Interval, PI checks whether the test results are normal, abnormal, and clinically significant.
  by cohort and visit, present continuous variables with subject count, mean, standard deviation, median, minimum, and maximum. For categorical variables, provide shift table.
X-ray | Before administration of investigational product at Baseline and Week 4 and within 4 hours after completion of administration
  by cohort and visit, present continuous variables with subject count, mean, standard deviation, median, minimum, and maximum. For categorical variables, provide shift table.
Physical Examinations | Up to 24 weeks
  Number of participants with clinically significant abnormalities in Physical Examinations after EN001 administration.
  Based on general appearance, head, ears/eyes/nose/throat, cardiovascular, respiratory, abdomen, skin, lymph nodes, extremities, musculoskeletal and neurologic, PI checks whether the test results are normal, abnormal, and clinically significant.
  By cohort and visit, present continuous variables with subject count, mean, standard deviation, median, minimum, and maximum. For categorical variables, provide shift table.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea